CLINICAL TRIAL: NCT04665986
Title: A Study to Evaluate Navelbine in Combination With Trastuzumab Plus Pertuzumab in Patients With HER2 Positive Early Stage or Locally Advanced Breast Cancer in Neoadjuvant Treatment
Brief Title: Neoadjuvant Study of Navelbine in Patients With HER2 Positive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NHP
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHP (Experimental): Navelbine, Herceptin, Pertuzumab
  Interventions: Drug: Navelbine
- THP (Active Comparator): Docetaxel, Herceptin, Pertuzumab
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Navelbine — Navelbine 25mg/m2 on day 1 and 8, every 3 weeks
  Arms: NHP
Drug: Docetaxel — Docetaxel 90mg/m2 on day 1, every 3 weeks
  Arms: THP

SUMMARY:
This is a randomized, double-blind multicenter Phase III study for evaluating the efficacy of neoadjuvant Navelbine plus trastuzumab and Pertuzumab versus Docetaxel plus trastuzumab and Pertuzumab given as neoadjuvant treatment in HER2 positive early-stage or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Female patients, 18 years ≤ age ≤ 80 years； Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1 Histologically confirmed invasive breast cancer（early stage or locally advanced） HER2 positive (HER2+++ by IHC or FISH+) Known hormone receptor status. Cardiovascular: Baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO Signed informed consent form (ICF)

Exclusion Criteria:

Metastatic disease (Stage IV) or inflammatory breast cancer Previous or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin, Carcinoma in situ of the cervix.

Clinically relevant cardiovascular disease: Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110); Unable or unwilling to swallow tablets.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
pCR | Through study completion, an average of 1 year
  Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery.

SECONDARY OUTCOMES:
DFS | Following surgery until Year 3
  Disease-free Survival
DDFS | Following surgery until Year 3
  Distance Disease-free Survival
ORR | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months
  Objective Response Rate